CLINICAL TRIAL: NCT03842800
Title: Characterizing Clinical and Pharmacological Neuroimaging Biomarkers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1111009332
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy; Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASD Patients (Other): This arm consists of patients diagnosed with Autism Spectrum Disorder (ASD) that will receive an MRI.
  Interventions: Other: MRI
- Schizophrenic Patients (Other): This arm consists of patients diagnosed with Schizophrenia that will receive an MRI.
  Interventions: Other: MRI
- Healthy Controls (Other): This arm consists of healthy control volunteer participants that will receive an MRI.
  Interventions: Other: MRI
- Healthy Controls with Ketamine (Experimental): This arm consists of healthy control volunteer participants that elect to receive ketamine prior to receiving an MRI.
  Interventions: Other: MRI; Drug: Ketamine

INTERVENTIONS:
Other: MRI — Patients and volunteers will receive an MRI.
  Other Names: Magnetic Resonance Imaging
Drug: Ketamine — Ketamine will be administered to a subset of healthy controls that agree to receive the drug as part of receiving an MRI.
  Arms: Healthy Controls with Ketamine

SUMMARY:
This study is part of a larger overall study that seeks to characterize clinical and pharmacological neuroimaging biomarkers. The purpose of this registered protocol is understand the effect of emotion on cognitions by specifically examining the effect of reward processing on working memory in patients with schizophrenia.

DETAILED DESCRIPTION:
Cognition rarely occurs in the 'real world' in isolation, and typically occurs under emotional influences that may alter how cognition occurs. Understanding these motivational and cognitive interactions will help better assess mechanisms that underlie the cognitive and negative symptoms of schizophrenia.

To better understand the effect of emotion on cognitions, this study will examine the effect of reward processing on working memory in patients with schizophrenia. To this end, this will be a two-pronged approach.

The first prong, is to understand the neural mechanisms of incentivized spatial working memory processes. fMRI will be used and a paradigm will be employed that combines reward processing and working memory to understand how patients with schizophrenia recruit neural systems in response to rewarded working memory.

To further understand this, this study will compare the neural effects in patients with schizophrenia with patients with depression, another group of psychiatric patients who also suffer from cognitive and motivational deficits. Both of these groups suffer from cognitive and motivational deficits, yet the treatments and disease presentations differ.

It is hypothesized that the ways in which cognitive and motivational processes interact in the brain will have some similarities, but also differences, that distinguish the two psychiatric illnesses. As part of this aim, a group of typical, healthy adults subjects will be recruited as a control. A subset of healthy participants that passed the medical and psychiatric screen will be invited to participate in the ketamine portion of the study which will be completed during the MRI session.

ELIGIBILITY:
Inclusion Criteria:

* For BOTH Non-Healthy Controls and Healthy Controls:
* Right-handed as determined by the Edinburgh handedness questionnaire (Oldfield, 1971).
* Premorbid IQ>70 determined by WAIS similarities and matrix reasoning subtests; Any history indicating learning disability, mental retardation, or attention deficit disorder will exclude the subject from participation.
* Must speak or read English at least 8th grade level or higher and to complete study evaluations.
* Must have intact vision or vision that can be corrected by glasses or contact lenses (corrected 20 20/20).
* Must be able to tolerate enclosed spaces ** only if participating in MRI portion.
* Female subjects must be postmenopausal for a least 1 year, surgically sterile, or using a reliable method of contraception at screening. Reliable methods of contraception include double-barrier methods (e.g. condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, or hormonal birth control methods. Women with positive serum pregnancy results at screening or self-reporting of pregnancy will be excluded from the study. ** only if participating in MRI portion.
* Must be free of metallic foreign objects in body, such as aneurysm clips or pacemakers, or a questionable history of metallic fragments ** only if participating in MRI portion.
* For Non-Healthy Controls Participants:
* Adult patients from the community meeting diagnostic criteria for schizophrenia, schizoaffective disorder, psychosis at risk syndrome, Major Depressive Disorder or autism spectrum disorders.
* Young adults (16-21) who are at risk of developing schizophrenia (have "prodromal schizophrenia") may be involved in the study.

Exclusion Criteria:

* For Healthy Controls:
* Evidence or history of serious medical or physical conditions, including severe endocrine disorder (Cushing's, Lupus), heart disorder (past history of heart attacks, angina), or other major systemic medical conditions (kidney, MS, CP, blindness, serious physical disability).
* Neurological conditions that might confound the results, including past stroke, seizures, dementia, brain tumor, brain surgery, neurological disease, head injury, or severe concussion (lasting >2 minutes in their life).
* Individual not larger than 55" around shoulders and widest part of chest (approx. 250lb limit) ** only if participating in MRI portion.
* Any other condition that is contra-indicated for fMRI if selected to participate in fMRI portion as determined by the MRRC safety screen. ** only if participating in MRI portion.
* Meeting current diagnostic criteria for any DSM-IV Axis I psychiatric disorders, determined by SCID-NP / MINI interviews.
* First-degree relative with Axis I DSM-IV disorder.
* Regular use of psychoactive drugs including anxiolytics and antidepressants.
* Meeting current DSM-IV abuse and/or dependence diagnostic criteria for other substances, other than nicotine in the past 6 months as determined by SCID-NP / MINI interviews (excluding caffeine).
* For Non-Healthy Controls:
* Medical. Evidence or history of serious medical or physical conditions, including severe endocrine disorder (Cushing's, Lupus), heart disorder (past history of heart attacks, angina), or other major systemic medical conditions (kidney, MS, CP, blindness, serious physical disability).
* Neurological conditions that might confound the results, including past stroke, seizures, dementia, brain tumor, brain surgery, neurological disease, head injury, or severe concussion (lasting >2 minutes in your lifetime).
* Individual not larger than 55" around shoulders and widest part of chest (approx. 250lb limit) ** only if participating in MRI portion.
* Any other condition that is contra-indicated for fMRI if selected to participate in fMRI portion as determined by the MRRC safety screen. ** only if participating in MRI portion.
* Meeting current diagnostic criteria for primary DSM-IV anxiety, depression or ADHD, determined by SCID-NP / MINI interview due to possible effects on cognition.
* Medication change within the past 2 weeks to avoid transient effects of medication regiment change; medication type and dose will be carefully recorded and used as a covariate in all analyses. Of note, if patients are not on medication (but are clinically stable) they will be invited to participate.
* History of any substance dependence disorder meeting DSM-IV criteria with the exception of nicotine and caffeine in the past 6 months. Meeting DSM-IV abuse and/or dependence diagnostic criteria for other substances in the past 6 months as determined by SCID / MINI interviews (again excluding caffeine and nicotine). Study will exclude for Specific Patterns of Substance Use. In addition, the study will exclude for use of stimulants, alcohol or heavy continued substance use defined as at least 3+ days per week for the duration of the last 6 months. In particular, we will not exclude for sporadic use of cannabis (defined as 3 or fewer marijuana cigarettes per week). Also, the study will exclude if a participant reports heavy habitual marijuana use, which we define more than 3 marijuana cigarettes per week over at least 90% of the weeks during a period of 6 months or more. Patterns of drug class, use pattern, frequency and history as well as the urine toxicology on the day of the assessment as well as all longitudinal followups will be assessed.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Working Memory (WM) | Up to 2 hours
  The tool used to measure working memory (WM) is a spatial working memory task. We measure angular accuracy of spatial working memory, and better accuracy is indicated by a lower angular distance. Subjects are asked to centrally fixate, and a circle appears on the screen briefly, and then disappears. Afterwards they see a gray circle that is linked to a joystick and are asked to move the gray circle to where they best remembered the initial circle to be. We care about the angular distance between where the initial circle appeared and where they placed the gray circle. The low range is 0 degrees, and the high range is 180 degrees. Scores are presented as averages and standard deviations.

SECONDARY OUTCOMES:
Behavior | Up to 2 hours
  The tool used to measure behavior is a spatial working memory task. We measure angular accuracy of spatial working memory, and better accuracy is indicated by a lower angular distance. We expect that patients with schizophrenia would have higher angular distances (ie, worse accuracy) than healthy control subjects on placebo, and patients with ASD. We expect that HCS on ketamine would have higher angular distances (ie worse accuracy), compared to when they are not on ketamine, and that this would approach the performance of patients with SCZ. The low range is 0 degrees, and the high range is 180 degrees. Scores are presented as averages and standard deviations.
BOLD | Up to 2 hours
  Regional BOLD (blood oxygen dependent) signal in the dorsolateral prefrontal cortex and parietal cortex. BOLD signal refers to the blood oxygen level dependent signal change measured using functional magnetic resonance imaging. It is an indirect marker of neural activity. The time series of BOLD signal changes is entered into a general linear model with our events of interest (WM maintenance) and we do statistics on the resulting beta weights.
Whole brain connectivity | Up to 2 hours
  Whole-brain connectivity refers to the correlation in time series between voxels. These analysis will specifically focus on the delay period subjects are maintaining a spatial location.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Anticevic, PhD, Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Magnetic Resonance Research Center, New Haven, Connecticut, United States